CLINICAL TRIAL: NCT05369221
Title: Feasibility of ReSpace™ Hydrogel to Establish a Stable Cervical-rectal Space
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Reunion Biotech Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN-CT-001-1
Record Dates: First submitted 2022-04-10; First posted 2022-05-11 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical Cancer; hydrogel spacer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReSpace™ (Experimental): The subjects who meet all the inclusion criteria and do not meet any of the exclusion criteria will be enrolled in this study. Subjects will undergo placement of ReSpace™ hydrogel.
  Interventions: Device: ReSpace™

INTERVENTIONS:
Device: ReSpace™ — All of the subjects will be injected with ReSpace™ hydrogel.

SUMMARY:
In this study, 5 subjects will be enrolled and the cumulative D2cc dose for rectum during brachytherapy will be recorded as the primary outcome measures.

DETAILED DESCRIPTION:
This is a phase I prospective study of 5 patients to determine if PEG hydrogel (ReSpace™) reduces the radiation dose delivered to the rectum during radiation therapy for cervical cancer by increasing the space between the cervix and the anterior rectal wall. In the other word, the purpose of this study is to assess whether the use of ReSpace™ hydrogel results in a reduction of radiation exposure to the anterior rectum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed cervical cancer who must be scheduled to undergo radical radiotherapy by means of intensity-modulated radiotherapy combined with 3D brachytherapy.
* Karnofsky score ≥ 70.
* Subjects aged ≥ 18 years and ≤ 75 years.
* Subjects must be able to cooperate in completing the entire study.
* The subjects' pelvic and abdominal cavity and joints are free of metal implants and can tolerate MRI.
* No contraindications to CT scanning.
* Subjects must be able to understand the purpose of the trial, voluntarily participate and sign an informed consent form.

Exclusion Criteria:

* Subjects who have received prior pelvic radiotherapy.
* Subjects whose target tumors have been previously treated (chemotherapy, immunotherapy, surgical treatment, etc.)
* Subjects with other primary malignancies
* Subjects with contraindications to radiotherapy, as determined by the investigators
* Subjects with injection site infections.
* Subjects who are allergic to the ingredients of the device.
* Subjects whose tumors invade the injection site and affect the injection process and injection safety, as determined by the investigators
* Persons with severe mental illness, cognitive impairment and thinking disorders.
* Participants in other drug clinical trials or medical device clinical trials 1 month prior to screening
* Pregnant or lactating women or those who plan to get pregnant within the last six months
* Subjects who cannot be followed up as prescribed by the doctor
* Other conditions that, in the judgment of the investigator, make the subject unsuitable for enrollment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
The cumulative D2cc dose for rectum during brachytherapy | 21 days post index procedure
  The mean of the cumulative rectum D2cc dose during brachytherapy will be calculated for subjects. which will be used to validate the parameter selection for phase II sample size estimation.

SECONDARY OUTCOMES:
Implantation success rate of hydrogel spacer | during procedure
  The success rate of hydrogel spacer implantation will be evaluated by the investigator for subjects.
Evaluation of device performance of hydrogel spacer | during procedure
  The ease of use of the test device will be evaluated by the investigator on the day of Operation. The evaluation items are as follows：
  1. Whether the device is easy to assemble.
  2. Whether the process of positioning the needle is smooth and whether it is easy to position the needle.
  3. Whether the device is easy to inject and whether the injection process is smooth.
Injection volume of hydrogel spacer | during procedure
  Recording the amount of hydrogel spacer injected in the subjects,which will be used to evaluate the reasonableness of the injected dose of ReSpace™ when hydrogel is injected between the rectum and cervix in women undergoing radiation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] de Freitas AC, Gurgel AP, Chagas BS, Coimbra EC, do Amaral CM. Susceptibility to cervical cancer: an overview. Gynecol Oncol. 2012 Aug;126(2):304-11. doi: 10.1016/j.ygyno.2012.03.047. Epub 2012 Apr 4. PMID 22484226
- [Background] Peach MS, Moore J, Giles W, Trainor J, Long T, Moon N, Hylton JE, Showalter TN, Libby B. Development and preclinical testing of a novel biodegradable hydrogel vaginal packing technology for gynecologic high-dose-rate brachytherapy. J Contemp Brachytherapy. 2018 Aug;10(4):306-314. doi: 10.5114/jcb.2018.77952. Epub 2018 Aug 31. PMID 30237814
- [Background] Kashihara T, Murakami N, Tselis N, Kobayashi K, Tsuchida K, Shima S, Masui K, Yoshida K, Takahashi K, Inaba K, Umezawa R, Igaki H, Ito Y, Kato T, Uno T, Itami J. Hyaluronate gel injection for rectum dose reduction in gynecologic high-dose-rate brachytherapy: initial Japanese experience. J Radiat Res. 2019 Jul 1;60(4):501-508. doi: 10.1093/jrr/rrz016. PMID 31034570